CLINICAL TRIAL: NCT05268588
Title: Effectiveness of an mHealth Interactive Education and Social Support Intervention for Improving Postnatal Health
Brief Title: mHealth India Postnatal Health Intervention Effectiveness
Acronym: Kushal Maa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Indraprastha Institute of Information Technology Delhi (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Sangath (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P0555059; R01HD108510 (NIH)
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Health Knowledge, Attitudes, Practice; Post Partum Depression; Breastfeeding; Nutrition, Healthy
Keywords: mHealth; group care
MeSH Terms: conditions — Behavior; Depression, Postpartum; Breast Feeding

STUDY DESIGN:
Intervention Model Description: The mHealth education and social support intervention includes tailored weekly educational content via interactive voice recognition and an android application, a phone-based provider-moderated group discussion, a provider-moderated group text chat, and referral to care as needed. Individuals are enrolled into groups of 20, have two intervention sessions prenatally and then have weekly meetings through six months postpartum for a total of 26 sessions. This model will be tested against the standard of care (3 postnatal visits in the first 7 days postpartum).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The mHealth education and social support intervention includes tailored weekly educational content via interactive voice recognition and an android application, a phone-based provider-moderated group discussion, a provider-moderated group text chat, and referral to care as needed. Individuals are enrolled into groups of 20, have two intervention sessions prenatally and then have weekly meetings through six months postpartum for a total of 26 sessions.
  Interventions: Behavioral: MESSSSAGE intervention
- Control Arm (No Intervention): Standard postnatal care.

INTERVENTIONS:
Behavioral: MESSSSAGE intervention — group mHealth education and social support intervention
  Arms: Intervention Arm

SUMMARY:
The goal of this study is to assess the effectiveness of a culturally-tailored mobile interactive education and support group intervention to supplement standard postpartum care activities in comparison to standard care alone on health-related behaviors and health outcomes in a randomized controlled trial among 2100 postpartum Indian women living in 3 geographically diverse Indian states to estimate the impact on maternal and neonatal health-related knowledge, health-related behaviors, and health outcomes. The investigators also seek to characterize mechanisms of impact including knowledge, social support, self-efficacy, and behavior change, and determine the cost-effectiveness.

DETAILED DESCRIPTION:
Maternal and infant mortality remain high in Northern India, at 167 per 100,000 live births and 49 per 1,000 live births, respectively. Access to perinatal care is increasing, yet gaps in care access and quality persist, particularly in peri-urban and rural areas. Steep drops in the perinatal continuum of care occur postpartum, with only 64% of mothers and 24% of infants receiving postpartum care, despite continuing maternal and infant risk. Ensuring continuity of high quality perinatal care into the postpartum period is key for maternal and infant health outcomes.

Postpartum care and support have received less focus than other perinatal continuum of care indicators yet are important for optimizing maternal and neonatal health and wellbeing. Significant logistical, sociodemographic and sociocultural barriers impede postpartum care access in India including postpartum seclusion, women's limited mobility, and geography. To overcome these barriers and reduce women's postpartum isolation through social support, an international team of maternal and infant health researchers and clinicians developed and pilot-tested a culturally-tailored mobile interactive education and support group intervention to supplement standard postpartum care activities: Maa Shishu Swasthya Sahayak Samooh (maternal and child health support group: MeSSSSage). MeSSSSage uses a provider-moderated group approach to increase women's communication with providers, to refer them to in-person care, and to connect them with a virtual social support group. Participants are recruited in late pregnancy and have 26 education and support sessions via audioconference facilitated by community health workers (two prenatal and weekly postpartum sessions through six months), plus engage in a text chat group. Group-based mHealth models are low cost and likely to be cost-effective. The participants overcome logistical and sociocultural barriers to postnatal care, and the participants have high acceptability and efficiency when used for other health issues. The pilot study results indicated high acceptability and feasibility and suggest preliminary effectiveness on maternal knowledge of best practices for facilitating postpartum health. Understanding intervention effectiveness on maternal health behaviors, key intervention pathways, and cost-effectiveness will inform the scalability of this intervention, with the potential to inform other similar ones.

The goal of this study is to assess the effectiveness of the 8-month MeSSSSage intervention in comparison to standard care alone on health-related behaviors and health outcomes in a fully powered randomized study, to test the conceptual model through analyzing the intervention's mechanisms of impact, and to determine cost-effectiveness. The investigators propose a randomized controlled trial (RCT) among 2100 postpartum Indian women living in 3 geographically diverse Indian states to estimate the impact of MeSSSSage on maternal and neonatal health-related knowledge, health-related behaviors, and health outcomes. The specific aims are to:

Aim 1: Estimate the effectiveness of a mobile interactive education and support group intervention (MeSSSSage) on postpartum behaviors for optimizing maternal and neonatal health in India. Within the 8-month RCT, the investigators will test the impact of the MeSSSSage intervention compared to standard care within 2100 Indian women. The primary effectiveness outcomes are exclusive breastfeeding, met need for postpartum contraceptives, and postpartum mental health. Secondary outcomes will incorporate additional maternal health behaviors and maternal and neonatal outcomes (e.g., appropriate care-seeking for illness, etc. see Table 2).

Aim 2: Characterize the mechanisms of impact of a mobile interactive education and support group intervention (MeSSSSage) on maternal and neonatal health in India. Within this RCT, the investigators will delineate the specific pathways through which the MeSSSSage intervention operates, including knowledge, social support, self-efficacy, and behavior change. The investigators will conduct mediation analyses using modern structural equation modeling and causal inference methods to identify the main drivers of the intervention impact to inform scalability.

Aim 3: Determine the cost-effectiveness of a mobile interactive education and support group intervention (MeSSSSage) in improving postpartum maternal and neonatal health as compared to the standard of care. The investigators will conduct cost analyses to determine intervention and standard of care costs, paying special attention to the value of social network belonging, and calculating opportunity cost. The investigators will conduct cost-effectiveness analysis (CEA) overall and stratified by social connectedness level to estimate the incremental cost-effectiveness ratio (ICER) of MeSSSSage in increasing exclusive breastfeeding, met need for postpartum contraception, and reducing postpartum depression, as compared to standard of care.

Perinatal educational and social support interventions are important for both physical and emotional well-being. The investigators anticipate that supplementing women's perinatal care within the postnatal period through an intervention approach that overcomes prevalent logistical and sociocultural challenges to care access through mHealth will have tangible impacts on the health and well-being of new mothers and infants. Estimating the impact of a mobile group intervention on maternal and infant health will inform scale-up of this accessible, acceptable, and feasible intervention among perinatal South Asian women, and can broadly inform the optimization of perinatal group care models for ensuring continuity across the full continuum of care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant (28-32 weeks gestational age)
* Speak local language
* Personal mobile phone or willing to accept study phone
* Able to provide informed consent

Exclusion Criteria:

* Do not speak local language
* No personal phone or unwilling to accept study phone
* Unable to provide informed consent

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2100 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding | 6 months
  Proportion of participants reporting exclusive breastfeeding at 3 and 6 months
Postpartum depression | 6 months
  Proportion of participants reporting postpartum depression symptoms at 3 and 6 months
Postpartum family planning adoption | 6 months
  Proportion of participants not wanting to become pregnant immediately having started a modern contraceptive method within 6 months postpartum

SECONDARY OUTCOMES:
Maternal and neonatal danger sign knowledge | 6 months
  Proportion of participants correctly identifying all maternal and neonatal danger signs by 6 months
Maternal and neonatal health care use | 6 months
  Proportion of participants seeking healthcare for maternal and neonatal concerns within 6 months
Neonatal preventive health care use | 6 months
  Proportion of participants having achieved target neonatal preventive care visits within 6 months
Infant vaccination | 6 months
  Proportion of participants having achieved recommended childhood vaccination schedule by 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alison M El Ayadi, ScD, Principal Investigator — University of California, San Francisco; Nadia G Diamond-Smith, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- India (3):
  - Post-Graduate Institute for Medical Education and Research, Chandīgarh, Haryana
  - Sangath, Bhopal, Madhya Pradesh
  - Indraprastha Institute for Information Technology, New Delhi, National Capital Territory of Delhi

IPD SHARING:
Plan to Share IPD: Yes
After study completion, de-identified data will be made available to other researchers upon reasonable request and completion of a data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: On study completion
Access Criteria: Request of study team.

REFERENCES:
- [Derived] El Ayadi AM, Duggal M, Gopalakrishnan L, Bagga R, Singh P, Lin T, Bhan A, Saunik S, Verma GS, Ahuja A, Kaur J, Tugnawat D, Gujarathi S, Singh A, Khan A, Chandke D, Dhir SK, Dhakne-Palwe S, Kumar P, Patil M, Kumar S, Vasaikar N, Weil L, Diamond-Smith N. Effectiveness of Kushal Maa, a group-based mhealth interactive education and social support intervention for maternal and neonatal health outcomes: study protocol for a multisite randomised controlled trial in India. BMJ Open. 2025 Jun 27;15(6):e104213. doi: 10.1136/bmjopen-2025-104213. PMID 40578858